CLINICAL TRIAL: NCT00284349
Title: Study to Investigate the Added Value of a Rehabilitation Brace in the Treatment at Home After a Fracture of the Ankle
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: René Verdonk, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/043
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Fracture of the Ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Use of a rehabilitation brace instead of a plaster

SUMMARY:
Comparison between immobilisation by a plaster and a rehabilitation brace for the treatment of a fracture of the ankle

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the ankle

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mobility of the ankle

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be